CLINICAL TRIAL: NCT02468193
Title: A Phase II, Open-label, Dose Titration, Multi-center Study to Assess the Safety/Tolerability and Efficacy of Osilodrostat in Patients With All Types of Endogenous Cushing's Syndrome Except Cushing's Disease
Brief Title: Study of Efficacy and Safety of Osilodrostat in Cushing's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C1201
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Cushing's Syndrome; Ectopic Corticotropin Syndrome; Adrenal Adenoma; Adrenal Carcinoma; AIMAH; PPNAD
Keywords: Cushing's syndrome; osilodrostat; LCI699; ectopic corticotropin syndrome; adrenal adenoma; adrenal carcinoma; ACTH-Independent Macronodular Adrenal Hyperplasia; AIMAH; Primary Pigmented Nodular Adrenal Dysplasia; PPNAD
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic; Adrenal Cortex Neoplasms; Acth-Independent Macronodular Adrenal Hyperplasia | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osilodrostat (Experimental): Patients in this arm took the study drug, osilodrostat.
  Interventions: Drug: Osilodrostat

INTERVENTIONS:
Drug: Osilodrostat — Osirodrostat 1mg, 5mg & 10mg in the form of film-coated tablets was used for oral administration.
  Other Names: LCI699

SUMMARY:
The study aim was to investigate the efficacy and safety of Osilodrostat in patients with Cushing's syndrome due to causes other than Cushing's disease in Japan.

DETAILED DESCRIPTION:
This was a Phase II, single arm, open-label, dose titration, multi-center study which consisted of two distinct Study Periods plus an optional extension period in non-CD patients with CS. The 3 Study Periods (two distinct Study Periods plus an optional extension period) were as follows:

Study Period I [Week 0 (Day 1) to Week-12]: Study Period I was the dose titration period to achieve a stable therapeutic dose and to assess the efficacy and safety of osilodrostat.

The dosing regimen of osilodrostat in this study was titrated according to the following escalation sequence: osilodrostat 2 mg bid, 5 mg bid, 10 mg bid, 20 mg bid, and 30 mg bid. Dose adjustments were based on the serum cortisol values measured by the local lab at each site. Osilodrostat titration was done weekly for the initial 4-weeks, up to a maximum dose of 10 mg bid.

The mean of three 24-hour UFC (mUFC) values were measured to evaluate the efficacy in this period.

Study Period II (After Week-12 to Week-48): Study Period II was the period to assess the sustainability of efficacy and long term safety.

During Study Period II, only patients who tolerated and agreed to continue osilodrostat treatment continued on the study. The patient was administered with the stable therapeutic dose which was achieved in the Study Period I.

Optional extension period (After Week-48): Patients who continued to receive clinical benefit, as assessed by the study Investigator and who wished to enter the extension period were reconsented at Week-48. Patients who entered the extension period continued to be treated with the study drug without interruption to be assessed for efficacy and safety. Patients who continued to benefit from study treatment as assessed by the study investigator and who completed Week-72 were offered to participate in a separate long-term safety follow-up study. The optional extension period ended after all patients had completed Week-72 or had discontinued early.

Post-treatment Follow-up: All patients had 30 days safety follow-up after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Cushing's syndrome [i.e. ectopic corticotropin syndrome, adrenal adenoma, adrenal carcinoma, ACTH-Independent Macronodular Adrenal Hyperplasia (AIMAH), or Primary Pigmented Nodular Adrenal Dysplasia (PPNAD)]
* For patients on medical treatment for hypercortisolism due to Cushing's syndrome, the washout periods had to be completed prior to baseline efficacy assessments

Exclusion Criteria:

* Patients with Cushing's disease
* History of hypersensitivity to osilodrostat or to drugs of similar chemical classes
* History of malignancy of any organ system, treated or untreated, within the past 5 years
* Patients receiving treatment for within 4 weeks or ≤5 x half-life of the agent (whichever is longer) before first dose of osilodrostat
* Patients with risk factors for QTc prolongation or Torsade de Pointes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (4):
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Chiba

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned subjects: 10 subjects Actual enrolled: 9 subjects
Pre-assignment Details: Planned subjects: 10 subjects
Period: Overall Study
Arm/Group | Osilodrostat
Started | 9
Completed Week-12 (Study Period I) | 7
Discontinued at or Prior to Week-12 | 2
Completed Week-12, Did Not Enter Per. II | 3
Completed Week-12, Entered Study Per. II | 4
Completed Week-48 (Study Period II) | 2
Discontinued at or Prior to Week48 | 2
Compl. Wk-48, Didn't Enter Opt. Ext. Per | 0
Compl. Wk-48, Entered Opt. Ext. Period | 2
Completed Optional Extension Period | 0
Discontinued Study in Optional Ext. Per. | 2
Completed | 3
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Subject/ Guardian decision | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Arm/Group | Osilodrostat
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (18.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 9
Type of disease [Number; unit: Participants]
  ACTH-Independent Macronodular Adrena;l Hyperplasia | 1
  Adrenal Adenoma | 5
  Ectopic Corticotropin Syndrome | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Mean Urine Free Cortisol (mUFC) at the Individual Level at Week 12
Description: Percent change from baseline in the mUFC at the individual patient level
Time Frame: Baseline, 12 weeks
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH- Patient 1 (n=1): number analyzed (Participants) | 1
  AIMAH- Patient 1 (n=1) | -99.0
  Adrenal adenoma - Patient 1 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma - Patient 1 (n=1) | -97.8
  Adrenal adenoma - Patient 2 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma - Patient 2 (n=1) | -94.5
  Adrenal adenoma - Patient 3 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma - Patient 3 (n=1) | -91.5
  Adrenal adenoma - Patient 4 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma - Patient 4 (n=1) | -81.8
  Adrenal adenoma - Patient 5 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma - Patient 5 (n=1) | -52.6
  Ectopic corticotropin syndrome - Patient 1 (n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome - Patient 1 (n=1) | -99.0
  Ectopic c orticotropin syndrome - Patient 2(n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome - Patient 3 (n=0): number analyzed (Participants) | 0

2. Secondary Outcome: Percent Change From Baseline in the mUFC at Individual Patient Level at Week 24 (Day 169) and Week 48 (Day 337)
Description: Percent change from baseline in the mUFC at the individual patient level
Time Frame: Baseline, Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt) 1: Week (Wk) 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1: Week (Wk) 24 (n=1) | -99.5
  AIMAH-Patient 1:Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient 1:Wk 48 (n=1) | -99.1
  Adrenal adenoma-Patient 1: Wk 24(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 1: Wk 48(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 2: Wk 24(n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 24(n=1) | -85.2
  Adrenal adenoma-Patient 2: Wk 48(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 24(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 48(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 24(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 48(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 24(n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 48(n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 1: Wk 24(n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 24(n=1) | -91.6
  Ectopic corticotropin syndrome-Pt 1: Wk 48(n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 48(n=1) | -91.0
  Ectopic corticotropin syndrome-Pt 2: Wk 24(n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 48(n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 24(n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 48(n=0): number analyzed (Participants) | 0

3. Secondary Outcome: Absolute Change From Baseline in the mUFC at Week 12 (Day 85), Week 24 (Day 169) and Week 48 (Day 337)
Description: Absolute change from baseline in the mUFC
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Median (Full Range); unit: nmol/24hr
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
nmol/24hr
  Week 12 (day 85)( n = 7) | -422.10 [-10487.5 to -157.0]
  Week 24 (day 169) (n = 3): number analyzed (Participants) | 3
  Week 24 (day 169) (n = 3) | -7428.10 [-9702.0 to -367.9]
  Week 48 (day 337) (n = 2): number analyzed (Participants) | 2
  Week 48 (day 337) (n = 2) | -8521.00 [-9640.5 to -7401.5]

4. Secondary Outcome: Percentage Change From Baseline in the mUFC at Week 12 (Day 85), Week 24 (Day 169) and Week 48 (Day 337)
Description: Percent change from baseline in the mUFC
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Median (Full Range); unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  Week 12 (day 85)( n = 7) | -94.47 [-99.0 to -52.6]
  Week 24 (day 169) (n = 3): number analyzed (Participants) | 3
  Week 24 (day 169) (n = 3) | -91.57 [-99.5 to -85.2]
  Week 48 (day 337) (n = 2): number analyzed (Participants) | 2
  Week 48 (day 337) (n = 2) | -95.04 [-99.1 to -91.0]

5. Secondary Outcome: Percentage of Participants With mUFC Response of Complete, Partial, and Overall Response
Description: Complete response rate = percentage of participants who had mUFC≤ ULN; Partial response rate = Percentage of participants who had mUFC>ULN and at least 50% reduction from baseline in mUFC. Overall response rate = Percentage of participants who had mUFC ≤ ULN or at least 50% reduction from baseline.
Time Frame: 12, 24 and 48 weeks
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osilodrostat
Number analyzed (Participants) | 9
Percentage of participants
  Week 12: Complete responders | 66.7 [29.9 to 92.5]
  Week 12: Partial responders | 11.1 [0.3 to 48.2]
  Week 12: Overall responders | 77.8 [40.0 to 97.2]
  Week 24: Complete responders (n =3): number analyzed (Participants) | 3
  Week 24: Complete responders (n =3) | 66.7 [9.4 to 99.2]
  Week 24: Partial responders (n = 3): number analyzed (Participants) | 3
  Week 24: Partial responders (n = 3) | 33.3 [0.8 to 90.6]
  Week 24: Overall responders (n = 3): number analyzed (Participants) | 3
  Week 24: Overall responders (n = 3) | 100 [29.2 to 100.0]
  Week 48: Complete responders (n = 2): number analyzed (Participants) | 2
  Week 48: Complete responders (n = 2) | 50.0 [1.3 to 98.7]
  Week 48: Partial responders (n = 2): number analyzed (Participants) | 2
  Week 48: Partial responders (n = 2) | 50.0 [1.3 to 98.7]
  Week 48: Overall responders (n = 2): number analyzed (Participants) | 2
  Week 48: Overall responders (n = 2) | 100 [15.8 to 100.0]

6. Secondary Outcome: Absolute Change From Baseline in Morning Serum Cortisol at Individual Level
Description: Absolute change from baseline in morning serum cortisol at the individual patient level
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: nmol/L
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
nmol/L
  AIMAH-Patient (Pt) 1: Week (Wk) 12 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1: Week (Wk) 12 (n = 1) | -607
  AIMAH-Patient 1: Wk 24 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 24 (n = 1) | -571
  AIMAH-Patient 1: Wk 48 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 48 (n = 1) | -580
  Adrenal adenoma-Patient 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 1: Wk 12 (n =1) | -334
  Adrenal adenoma-Patient 1:Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 1: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 2: Wk 12(n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 12(n =1) | -157
  Adrenal adenoma-Patient 2: Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 24 (n =1) | -135
  Adrenal adenoma-Patient 2: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 3: Wk 12 (n =1) | -300
  Adrenal adenoma-Patient 3: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 4: Wk 12 (n =1) | -30
  Adrenal adenoma-Patient 4: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 5: Wk 12 (n =1) | -13
  Adrenal adenoma-Patient 5: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1) | -949
  Ectopic corticotropin syndrome-Pt 1: Wk24 (n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk24 (n=1) | -927
  Ectopic corticotropin syndrome-Pt 1: Wk48 (n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk48 (n=1) | -861
  Ectopic corticotropin syndrome-Pt 2: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk48 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk24 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk48 (n=0): number analyzed (Participants) | 0

7. Secondary Outcome: Percentage Change From Baseline in Morning Serum Cortisol at Individual Level
Description: Percentage change from baseline in morning serum cortisol at the individual patient level
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt) 1: Week (Wk) 12 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1: Week (Wk) 12 (n = 1) | -73.3
  AIMAH-Patient 1: Wk 24 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 24 (n = 1) | -69.0
  AIMAH-Patient 1: Wk 48 (n = 1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 48 (n = 1) | -70.0
  Adrenal adenoma-Patient 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 1: Wk 12 (n =1) | -78.0
  Adrenal adenoma-Patient 1:Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 1: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 2: Wk 12(n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 12(n =1) | -50.8
  Adrenal adenoma-Patient 2: Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 24 (n =1) | -43.7
  Adrenal adenoma-Patient 2: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 3: Wk 12 (n =1) | -56.1
  Adrenal adenoma-Patient 3: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 4: Wk 12 (n =1) | -8.7
  Adrenal adenoma-Patient 4: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 5: Wk 12 (n =1) | -3.5
  Adrenal adenoma-Patient 5: Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1) | -71.4
  Ectopic corticotropin syndrome-Pt 1: Wk24 (n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk24 (n=1) | -69.7
  Ectopic corticotropin syndrome-Pt 1: Wk48 (n=1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk48 (n=1) | -64.7
  Ectopic corticotropin syndrome-Pt 2: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk24 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk48 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk24 (n=0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk48 (n=0): number analyzed (Participants) | 0

8. Secondary Outcome: Absolute Change From Baseline in ACTH and Other Adrenal Steroid Hormones at Individual Level
Description: Absolute change from baseline in several steroid hormones at individual levels: ACTH, Serum 11-deoxycorticosterone, Aldosterone, Estradiol
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: pmol/L
Groups:
- ACTH: Adrenocorticotropic hormone
- Serum 11-deoxycorticosterone: adrenal steroid hormones: Serum 11-deoxycorticosterone
- Aldosterone: adrenal steroid hormones: Aldosterone
- Estradiol: adrenal steroid hormones: Estradiol
Arm/Group | ACTH | Serum 11-deoxycorticosterone | Aldosterone | Estradiol
Number analyzed (Participants) | 7 | 7 | 7 | 7
pmol/L
  AIMAH-Patient (Pt) 1 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n=1,1,1,1) | 0 | 2179 | 52 | 705
  AIMAH-Pt 1 Wk 24 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 24 (n=1,1,1,1) | 0 | 3601 | 236 | 235
  AIMAH-Pt 1 Wk 48 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 48 (n=1,1,1,1) | 0 | 454 | 170 | 400
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1,1,1) | 1.1 | 2966 | -27 | -404
  Adrenal adenoma-Pt 1 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1,1,1) | 0 | 5145 | -981 | 4
  Adrenal adenoma-Pt 2 Wk 24(n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24(n=1,1,1,1) | 0 | 0 | 450 | -4
  Adrenal adenoma-Pt 2 Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1,1,1) | 0 | 0 | -147 | 77
  Adrenal adenoma-Pt 3 Wk 24 (n=0, 0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48(n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1,1,1) | 0 | 787 | 3 | 18
  Adrenal adenoma-Pt 4 Wk 24 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1,1,1) | 0 | 0 | 0 | -11
  Adrenal adenoma-Pt 5 Wk 24 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 1: Wk 12 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 12 (n=1,1,1,1) | -67.7 | -696 | 145 | 51
  Ectopic ACTH syndrome-Pt 1: Wk 24 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 24 (n=1,1,1,1) | -47.3 | -91 | 40 | -11
  Ectopic ACTH syndrome-Pt 1: Wk 48 (n=1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 48 (n=1,1,1,1) | 13.3 | -91 | 37 | 11
  Ectopic ACTH syndrome-Pt 2: Wk 12 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2: Wk 24 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2: Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3: Wk 12 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3: Wk 24 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3: Wk 48 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage Change From Baseline in ACTH and Other Adrenal Steroid Hormones at Individual Level
Description: Percent change from baseline in several steroid hormones at individual levels: ACTH, Serum 11-deoxycorticosterone, Aldosterone, Estradiol
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | ACTH | Serum 11-deoxycorticosterone | Aldosterone | Estradiol
Number analyzed (Participants) | 7 | 7 | 7 | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n =0,1,0,1): number analyzed (Participants) | 0 | 1 | 0 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =0,1,0,1) |  | 118.0 |  | 1282
  AIMAH-Pt 1 Wk 24 (n=0,1,0,1): number analyzed (Participants) | 0 | 1 | 0 | 1
  AIMAH-Pt 1 Wk 24 (n=0,1,0,1) |  | 195.1 |  | 427.3
  AIMAH-Pt 1 Wk 48 (n=0,1,0,1): number analyzed (Participants) | 0 | 1 | 0 | 1
  AIMAH-Pt 1 Wk 48 (n=0,1,0,1) |  | 24.6 |  | 727.3
  Adrenal adenoma-Pt 1 Wk 12 (n =0,0,1,1): number analyzed (Participants) | 0 | 0 | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =0,0,1,1) |  |  | -13.9 | -53.7
  Adrenal adenoma-Pt 1 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =0,0,1,1): number analyzed (Participants) | 0 | 0 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =0,0,1,1) |  |  | -100 | 1.9
  Adrenal adenoma-Pt 2 Wk 24 (n =0,0,1,1): number analyzed (Participants) | 0 | 0 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =0,0,1,1) |  |  | 45.9 | -1.9
  Adrenal adenoma-Pt 2 Wk 48 (n =0,0,0, 0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =0,0,1,1): number analyzed (Participants) | 0 | 0 | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =0,0,1,1) |  |  | -75.0 | 513.3
  Adrenal adenoma-Pt 3 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =0,0,1,1): number analyzed (Participants) | 0 | 0 | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =0,0,1,1) |  |  | 10.0 | 120.0
  Adrenal adenoma-Pt 4 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =0,0,0,1): number analyzed (Participants) | 0 | 0 | 0 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =0,0,0,1) |  |  |  | -100
  Adrenal adenoma-Pt 5 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 1: Wk 12 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 12 (n=1,1,0,1) | -71.6 | -100 |  | 72.9
  Ectopic ACTH syndrome-Pt 1: Wk 24 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 24 (n=1,1,0,1) | -50.0 | -13.1 |  | -15.7
  Ectopic ACTH syndrome-Pt 1: Wk 48 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Ectopic ACTH syndrome-Pt 1: Wk 48 (n=1,1,0,1) | 14.1 | -13.1 |  | 15.7
  Ectopic ACTH syndrome-Pt 2: Wk 12 (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Absolute Change From Baseline in Other Adrenal Steroid Hormones at Individual Levels
Description: Absolute change from baseline in several steroid hormones at individual levels: Serum 11-deoxycortisol, Testosterone
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: nmol/L
Groups:
- Serum 11-deoxycortisol: adrenal steroid hormones: Serum 11-deoxycortisol
- Testosterone: adrenal steroid hormones: Testosterone
Arm/Group | Serum 11-deoxycortisol | Testosterone
Number analyzed (Participants) | 7 | 7
nmol/L
  AIMAH-Patient (Pt) 1 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n = 1,1) | -4.35 | 0.76
  AIMAH-Pt 1 Wk 24 (n = 1,1): number analyzed (Participants) | 1 | 1
  AIMAH-Pt 1 Wk 24 (n = 1,1) | -8.5 | 0.66
  AIMAH-Pt 1 Wk 48 (n = 1,1): number analyzed (Participants) | 1 | 1
  AIMAH-Pt 1 Wk 48 (n = 1,1) | -15.54 | -0.03
  Adrenal adenoma-Pt 1 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n = 1,1) | 6.91 | 0.31
  Adrenal adenoma-Pt 1 Wk 24 (n =0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n = 1,1) | 2.81 | 0.11
  Adrenal adenoma-Pt 2 Wk 24 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n = 1,1) | -0.64 | -0.35
  Adrenal adenoma-Pt 2 Wk 48 (n = 0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n = 1,1) | 7.34 | 0.42
  Adrenal adenoma-Pt 3 Wk 24 (n = 0, 0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n = 1,1) | 3.5 | 0.03
  Adrenal adenoma-Pt 4 Wk 24 (n = 0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n = 0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n = 1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n = 1,1) | -1.39 | 0
  Adrenal adenoma-Pt 5 Wk 24 (n =0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n = 0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n = 1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n = 1,1) | -15.81 | 5.83
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n = 1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n = 1,1) | -12.41 | -2.71
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n = 1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n = 1,1) | -2.52 | -2.01
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n = 0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n = 0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n = 0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n =0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n = 0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48(n = 0,0): number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage Change From Baseline in Other Adrenal Steroid Hormones at Individual Levels
Description: Percent change from baseline in several steroid hormones at individual levels: Serum 11-deoxycortisol, Testosterone
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Serum 11-deoxycortisol | Testosterone
Number analyzed (Participants) | 7 | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n=1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n=1, 1) | -17.8 | 73.1
  AIMAH-Pt 1 Wk 24 (n=1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Pt 1 Wk 24 (n=1, 1) | -34.9 | 63.5
  AIMAH-Pt 1 Wk 48 (n=1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Pt 1 Wk 48 (n=1, 1) | -63.7 | -2.9
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1) | 143.7 | 100.0
  Adrenal adenoma-Pt 1 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1) | 108.9 | 10.6
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1) | -24.8 | -33.7
  Adrenal adenoma-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1, 1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1, 1) | 127.2 | 93.3
  Adrenal adenoma-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0,0: number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1, 1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1, 1) | 267.2 | 14.3
  Adrenal adenoma-Pt 4 Wk 24 (n=0,0: number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0,0: number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1) | -43.2 | 0.0
  Adrenal adenoma-Pt 5 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1, 1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1, 1) | -64.8 | 96.5
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1, 1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1, 1) | -50.9 | -44.9
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1, 1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1, 1) | -10.3 | -33.3
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameter, Fasting Glucose, at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameter fasting glucose, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: mmol/L
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
mmol/L
  AIMAH-Patient (Pt) 1 Wk 12 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1) | -0.78
  AIMAH-Patient (Pt) 1 Wk 24 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 24 (n =1) | -0.84
  AIMAH-Patient (Pt) 1 Wk 48 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 48 (n =1) | -0.78
  Adrenal adenoma-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1) | 1.22
  Adrenal adenoma-Pt 1 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1) | -1.89
  Adrenal adenoma-Pt 2 Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1) | 0.22
  Adrenal adenoma-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1) | -0.28
  Adrenal adenoma-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1) | -0.67
  Adrenal adenoma-Pt 4 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1) | -0.05
  Adrenal adenoma-Pt 5 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n =1) | -0.33
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1) | -0.39
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1) | 0.06
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0

13. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameter, Fasting Glucose, at Individual Level
Description: Percentasge change in cardiovascular-related metabolic parameter fasting glucose, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1) | -15.3
  AIMAH-Patient (Pt) 1 Wk 24 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 24 (n =1) | -16.4
  AIMAH-Patient (Pt) 1 Wk 48 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 48 (n =1) | -15.3
  Adrenal adenoma-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1) | 24.2
  Adrenal adenoma-Pt 1 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1) | -27.2
  Adrenal adenoma-Pt 2 Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1) | 3.2
  Adrenal adenoma-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1) | -5.0
  Adrenal adenoma-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1) | -11.3
  Adrenal adenoma-Pt 4 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1) | -0.9
  Adrenal adenoma-Pt 5 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n =1) | -5.9
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1) | -7.0
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1) | 1.1
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0

14. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameter, HbA1c, at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameter HbA1c associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage of HbA1c
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage of HbA1c
  AIMAH-Patient (Pt) 1 Wk 12 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n=1) | -0.1
  AIMAH-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 24 (n=1) | -0.1
  AIMAH-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 48 (n=1) | -0.2
  Adrenal adenoma-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1) | 0.3
  Adrenal adenoma-Pt 1 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1) | -0.4
  Adrenal adenoma-Pt 2 Wk 24 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1) | -0.7
  Adrenal adenoma-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1) | -1.4
  Adrenal adenoma-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1) | -0.9
  Adrenal adenoma-Pt 4 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1) | -0.1
  Adrenal adenoma-Pt 5 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1) | 0.3
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1) | 0.5
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1) | 0.8
  Ectopic ACTH syndrome-Pt 2 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0

15. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameter, HbA1c, at Individual Level
Description: Percentage change in cardiovascular-related metabolic parameter HbA1c associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n=1) | -1.8
  AIMAH-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 24 (n=1) | -1.8
  AIMAH-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 48 (n=1) | -3.6
  Adrenal adenoma-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1) | 6.2
  Adrenal adenoma-Pt 1 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1) | -6.5
  Adrenal adenoma-Pt 2 Wk 24 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1) | -11.3
  Adrenal adenoma-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1) | -20.3
  Adrenal adenoma-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1) | -12.2
  Adrenal adenoma-Pt 4 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1) | -1.5
  Adrenal adenoma-Pt 5 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1) | 5.4
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1) | 8.9
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1) | 14.3
  Ectopic ACTH syndrome-Pt 2 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0

16. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameters, Cholesterol, HDL Cholesterol, LDL Cholesterol & Triglycerides, at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameters: cholesterol, HDL cholesterol, LDL cholesterol & triglycerides, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: mmol/L
Groups:
- Cholesterol; HDL Cholesterol; LDL Cholesterol; Triglycerides: Patients in this arm took the study drug, osilodrostat.
Arm/Group | Cholesterol | HDL Cholesterol | LDL Cholesterol | Triglycerides
Number analyzed (Participants) | 7 | 7 | 7 | 7
mmol/L
  AIMAH-Patient (Pt) 1 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1,1,1,1) | -0.67 | -0.85 | 0.21 | -0.87
  AIMAH-Pt 1 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 24 (n =1,1,1,1) | -0.65 | -1.01 | 0.18 | -0.64
  AIMAH-Pt 1 Wk 48 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 48 (n =1,1,1,1) | -0.72 | -0.57 | -0.08 | -0.76
  Adrenal adenoma-Pt 1 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1,1,1,1) | -1.56 | -0.26 | -1.11 | -1.42
  Adrenal adenoma-Pt 1 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1,1,1,1) | -0.54 | -0.64 | -0.26 | 0.11
  Adrenal adenoma-Pt 2 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1,1,1,1) | 0.26 | -0.33 | 0.31 | 0.08
  Adrenal adenoma-Pt 2 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1,1,1,1) | -0.55 | -0.16 | -0.19 | -1.36
  Adrenal adenoma-Pt 3 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1,1,1,1) | 1.09 | 0.18 | 0.72 | 0.58
  Adrenal adenoma-Pt 4 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1,1,1,1) | -0.39 | -0.21 | -0.18 | 0.44
  Adrenal adenoma-Pt 5 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1,1,1,1) | -0.16 | 0.16 | -0.11 | -0.47
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1,1,1,1) | -0.26 | 0.49 | -0.29 | -0.83
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1,1,1,1) | -0.08 | 0.29 | -0.31 | 0.22
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0,0,0,0,): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameters, Cholesterol, HDL Cholesterol, LDL Cholesterol & Triglycerides, at Individual Level
Description: Percent change in cardiovascular-related metabolic parameters: cholesterol, HDL cholesterol, LDL cholesterol & triglycerides, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Cholesterol | HDL Cholesterol | LDL Cholesterol | Triglycerides
Number analyzed (Participants) | 7 | 7 | 7 | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1,1,1,1) | -11.1 | -33.2 | 6.3 | -49.4
  AIMAH-Pt 1 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 24 (n =1,1,1,1) | -10.7 | -39.5 | 5.4 | -36.4
  AIMAH-Pt 1 Wk 48 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  AIMAH-Pt 1 Wk 48 (n =1,1,1,1) | -11.9 | -22.3 | -2.4 | -43.2
  Adrenal adenoma-Pt 1 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1,1,1,1) | -23.0 | -27.1 | -24.9 | -28.8
  Adrenal adenoma-Pt 1 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1,1,1,1) | -11.9 | -34.4 | -10.6 | 12.5
  Adrenal adenoma-Pt 2 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1,1,1,1) | 5.7 | -17.7 | 12.6 | 9.1
  Adrenal adenoma-Pt 2 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1,1,1,1) | -9.5 | -9.4 | -5.5 | -56.7
  Adrenal adenoma-Pt 3 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1,1,1,1) | 23.0 | 15.5 | 26.5 | 46.8
  Adrenal adenoma-Pt 4 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1,1,1,1) | -8.7 | -11.4 | -9.3 | 33.3
  Adrenal adenoma-Pt 5 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1,1,1,1) | -3.8 | 12.4 | -4.5 | -32.0
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1,1,1,1) | -6.2 | 38.0 | -11.8 | -56.5
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1,1,1,1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1,1,1,1) | -1.9 | 22.5 | -12.6 | 15.0
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameter, BMI, at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameter: BMI, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: kg/m^2
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
kg/m^2
  AIMAH-Patient (Pt) 1 Wk 12 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1) | -0.5
  AIMAH-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 24 (n =1) | -2.3
  AIMAH-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 48 (n =1) | -1.6
  Adrenal adenoma-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1) | 0.6
  Adrenal adenoma-Pt 1 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1) | -1.2
  Adrenal adenoma-Pt 2 Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1) | -3.6
  Adrenal adenoma-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1) | 0.7
  Adrenal adenoma-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1) | 0.2
  Adrenal adenoma-Pt 4 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1) | 0.1
  Adrenal adenoma-Pt 5 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1) | 1.8
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1) | 3.0
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1) | 3.6
  Ectopic ACTH syndrome-Pt 2 Wk 12(n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0

19. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameter, BMI, at Individual Level
Description: Percent change in cardiovascular-related metabolic parameter: BMI, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt) 1 Wk 12 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt) 1 Wk 12 (n =1) | -2.1
  AIMAH-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 24 (n =1) | -9.6
  AIMAH-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  AIMAH-Pt 1 Wk 48 (n =1) | -6.7
  Adrenal adenoma-Pt 1 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n =1) | 1.9
  Adrenal adenoma-Pt 1 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n =1) | -3.1
  Adrenal adenoma-Pt 2 Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n =1) | -9.4
  Adrenal adenoma-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n =1) | 3.3
  Adrenal adenoma-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n =1) | 0.9
  Adrenal adenoma-Pt 4 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n =1) | 0.5
  Adrenal adenoma-Pt 5 Wk 24 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n =1) | 7.4
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n =1) | 12.3
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n =1) | 14.8
  Ectopic ACTH syndrome-Pt 2 Wk 12(n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n =0): number analyzed (Participants) | 0

20. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameter, Waist Circumference, at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameter: Waist circumference, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: cm
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
cm
  AIMAH-Patient (Pt)1 Wk 12 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt)1 Wk 12 (n=1) | -2.0
  AIMAH-Pt1 Wk 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt1 Wk 24 (n=1) | -7.5
  AIMAH-Pt1 Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt1 Wk 48 (n=1) | -5.5
  Adrenal adenoma-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1) | -2.0
  Adrenal adenoma-Pt 1 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1) | -1.0
  Adrenal adenoma-Pt 2 Wk 24 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1) | -8.0
  Adrenal adenoma-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1) | -4.0
  Adrenal adenoma-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1) | 1.0
  Adrenal adenoma-Pt 4 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1) | -0.3
  Adrenal adenoma-Pt 5 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1) | 2.5
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1) | 11.0
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1) | 9.5
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0

21. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameter, Waist Circumference, at Individual Level
Description: Percent change in cardiovascular-related metabolic parameter: Waist circumference, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
percentage change
  AIMAH-Patient (Pt)1 Wk 12 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient (Pt)1 Wk 12 (n=1) | -2.4
  AIMAH-Pt1 Wk 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt1 Wk 24 (n=1) | -9.0
  AIMAH-Pt1 Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Pt1 Wk 48 (n=1) | -6.6
  Adrenal adenoma-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1) | -1.8
  Adrenal adenoma-Pt 1 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1) | -0.9
  Adrenal adenoma-Pt 2 Wk 24 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1) | -7.1
  Adrenal adenoma-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1) | -4.9
  Adrenal adenoma-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1) | 1.1
  Adrenal adenoma-Pt 4 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1) | -0.4
  Adrenal adenoma-Pt 5 Wk 24 (n=0): number analyzed (Participants) | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12 (n=1) | 2.9
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1) | 12.9
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1): number analyzed (Participants) | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1) | 11.1
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12(n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0): number analyzed (Participants) | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0): number analyzed (Participants) | 0

22. Secondary Outcome: Absolute Change From Baseline in Cardiovascular-related Metabolic Parameter, Sitting Blood Pressure (BP) at Individual Level
Description: Absolute change in cardiovascular-related metabolic parameter: sitting systolic BP & sitting diastolic BP, associated with Cushing's syndrome (CS)
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: mmHg
Groups:
- Sitting Systolic BP; Sitting Diastolic BP: Patients in this arm took the study drug, osilodrostat.
Arm/Group | Sitting Systolic BP | Sitting Diastolic BP
Number analyzed (Participants) | 7 | 7
mmHg
  AIMAH-Patient (Pt) 1Wk 12 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1Wk 12 (n =1, 1) | -44.3 | -31.0
  AIMAH-Patient (Pt) 1 Wk 24 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 24 (n =1, 1) | -48.34 | -32.66
  AIMAH-Patient (Pt) 1 Wk 48 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 48 (n =1, 1) | -40.34 | -19.0
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1) | 11.67 | -3.67
  Adrenal adenoma-Pt 1 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1) | -50.67 | -37.0
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1) | -32.33 | -26.66
  Adrenal adenoma-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1) | -16.0 | -6.67
  Adrenal adenoma-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1) | -6.67 | 7.33
  Adrenal adenoma-Pt 4 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1) | 11.0 | 3.33
  Adrenal adenoma-Pt 5 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n=1,1) | -17.67 | -13.67
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1,1) | 4.33 | 4.0
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1,1) | -1.0 | -0.67
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percentage Change From Baseline in Cardiovascular-related Metabolic Parameter, Sitting Blood Pressure (BP) at Individual Level
Description: Percentage change in cardiovascular-related metabolic parameter: sitting systolic BP & sitting diastolic BP, associated with Cushing's syndrome
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: percentage change
Arm/Group | Sitting Systolic BP | Sitting Diastolic BP
Number analyzed (Participants) | 7 | 7
percentage change
  AIMAH-Patient (Pt) 1Wk 12 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1Wk 12 (n =1, 1) | -31.1 | -32.5
  AIMAH-Patient (Pt) 1 Wk 24 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 24 (n =1, 1) | -33.9 | -34.3
  AIMAH-Patient (Pt) 1 Wk 48 (n =1, 1): number analyzed (Participants) | 1 | 1
  AIMAH-Patient (Pt) 1 Wk 48 (n =1, 1) | -28.3 | -19.9
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 1 Wk 12 (n=1,1) | 9.2 | -4.1
  Adrenal adenoma-Pt 1 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 1 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 12 (n=1,1) | -31.3 | -33.2
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 2 Wk 24 (n=1,1) | -20.0 | -23.9
  Adrenal adenoma-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 3 Wk 12 (n=1,1) | -12.3 | -8.9
  Adrenal adenoma-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 3 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 4 Wk 12 (n=1,1) | -4.3 | 9.9
  Adrenal adenoma-Pt 4 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 4 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1): number analyzed (Participants) | 1 | 1
  Adrenal adenoma-Pt 5 Wk 12 (n=1,1) | 9.3 | 5.1
  Adrenal adenoma-Pt 5 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Adrenal adenoma-Pt 5 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 1 Wk 12(n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 12(n=1,1) | -14.1 | -16.5
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 24 (n=1,1) | 3.4 | 4.8
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1,1): number analyzed (Participants) | 1 | 1
  Ectopic ACTH syndrome-Pt 1 Wk 48 (n=1,1) | -0.8 | -0.8
  Ectopic ACTH syndrome-Pt 2 Wk 12 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 2 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 12 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 24 (n=0,0): number analyzed (Participants) | 0 | 0
  Ectopic ACTH syndrome-Pt 3 Wk 48 (n=0,0): number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Total Scores in Patient-Reported Outcomes Health-related Quality of Life (QoL) as Assessed by Cushing QoL at Individual Level
Description: The Cushing's Disease Health-Related Quality of Life Questionnaire (Cushing QoL) (version 1.0) was developed to evaluate quality of life in patients with Cushing's syndrome (Webb et al 2008). The Cushing QoL is comprised of 12 items that capture patient responses on seven concepts: daily activities, healing and pain, mood and self-confidence, social concerns, physical appearance, memory and concern about the future. Each questionnaire of the Cushing QOL has a scale of 1-5 where '1' corresponding to 'Always' or 'Very much' and '5' to 'Never' or 'Not at all'. The lower the score, the greater the impact on HRQoL. The score is the sum of all the item response and can range from 12 (worst) to 60 points (best).
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: scores on a scale
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
scores on a scale
  AIMAH-Patient 1: Week (Wk) 12 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Week (Wk) 12 (n=1) | 48
  AIMAH-Patient 1: Wk 24 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 24 (n=1) | 51
  AIMAH-Patient 1: Wk 48 (n=1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 48 (n=1) | 47
  Adrenal adenoma-Patient 1: Wk 12(n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 1: Wk 12(n=1) | 29
  Adrenal adenoma-Patient 1: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 1: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 2: Wk 12(n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 12(n=1) | 18
  Adrenal adenoma-Patient 2: Wk 24 (n = 1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 24 (n = 1) | 22
  Adrenal adenoma-Patient 2: Wk 48 (n =0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 3: Wk 12 (n =1) | 29
  Adrenal adenoma-Patient 3: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 4: Wk 12 (n =1) | 38
  Adrenal adenoma-Patient 4: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 12 (n=1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 5: Wk 12 (n=1) | 45
  Adrenal adenoma-Patient 5: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 48 (n = 0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1) | 31
  Ectopic corticotropin syndrome-Pt 1: Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 24 (n =1) | 33
  Ectopic corticotropin syndrome-Pt 1: Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 48 (n =1) | 23
  Ectopic corticotropin syndrome-Pt 2: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 12 n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 48 (n =0): number analyzed (Participants) | 0

25. Secondary Outcome: Total Scores in Patient-Reported Outcomes Health-related Quality of Life (QoL) as Assessed by Beck Depression Inventory II (BDI-ll) Depression Score at Individual Level
Description: The Beck Depression Inventory II (BDI-II) is a patient reported instrument that consists of 21 items designed to assess the intensity of depression in clinical & normal patients in the preceding two weeks. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. Each of 21 items corresponds to a symptom of depression and the sum of total score will be calculated where each item has a four-point scale ranging from 0 to 3, leading to a total score from zero to 63.
Time Frame: Baseline, Week 12 (day 85), Week 24 (day 169) and Week 48 (day 337)
Population: Full Analysis Set (FAS): Comprised of all enrolled patients who received at least one dose of osilodrostat.
Measure: Number; unit: scores on a scale
Arm/Group | Osilodrostat
Number analyzed (Participants) | 7
scores on a scale
  AIMAH-Patient 1: Week (Wk) 12 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Week (Wk) 12 (n =1) | 4
  AIMAH-Patient 1: Wk 24 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 24 (n =1) | 15
  AIMAH-Patient 1: Wk 48 (n =1): number analyzed (Participants) | 1
  AIMAH-Patient 1: Wk 48 (n =1) | 12
  Adrenal adenoma-Patient 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 1: Wk 12 (n =1) | 33
  Adrenal adenoma-Patient 1: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 1: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 2: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 12 (n =1) | 35
  Adrenal adenoma-Patient 2: Wk 24 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 2: Wk 24 (n =1) | 37
  Adrenal adenoma-Patient 2: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 3: Wk 12 (n =1) | 30
  Adrenal adenoma-Patient 3: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 3: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 4: Wk 12 (n =1) | 26
  Adrenal adenoma-Patient 4: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 4: Wk 48 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 12 (n =1): number analyzed (Participants) | 1
  Adrenal adenoma-Patient 5: Wk 12 (n =1) | 10
  Adrenal adenoma-Patient 5: Wk 24 (n = 0): number analyzed (Participants) | 0
  Adrenal adenoma-Patient 5: Wk 48 (n = 0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 12 (n =1) | 9
  Ectopic corticotropin syndrome-Pt 1: Wk 24 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 24 (n =1) | 10
  Ectopic corticotropin syndrome-Pt 1: Wk 48 (n =1): number analyzed (Participants) | 1
  Ectopic corticotropin syndrome-Pt 1: Wk 48 (n =1) | 22
  Ectopic corticotropin syndrome-Pt 2: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 2: Wk 48 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 12 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 24 (n =0): number analyzed (Participants) | 0
  Ectopic corticotropin syndrome-Pt 3: Wk 48 (n =0): number analyzed (Participants) | 0

26. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 0
Description: Osilodrostat plasma concentration data at each time-point were summarized by incident dose. About a half of pre-dose concentration data were excluded from analysis due to deviation from the pre-defined acceptable time window.
Time Frame: Week 0
Population: Pharmacokinetic analysis set (PAS): Consisted of all patients who received at least one dose of osilodrostat and had at least one evaluable PK concentration at any visit (post-first-dose).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Osilodrostat 1mg: Patients in this arm took 1mg of study drug, osilodrostat.
- Osilodrostat 2mg: Patients in this arm took 2mg of study drug, osilodrostat.
- Osilodrostat 3mg: Patients in this arm took 3mg of study drug, osilodrostat.
- Osilodrostat 5mg: Patients in this arm took 5mg of study drug, osilodrostat.
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 1 | 8 | 0 | 0
ng/mL
  Week 0: 0.75 hour post-dose | 0.971 (NA) — N/A : not enough participants to calculate the standard deviation | 0.405 (0.673) |  |
  Week 0: 2 hours post-dose | 5.11 (NA) — N/A : not enough participants to calculate the standard deviation | 5.29 (4.94) |  |
  Week 0: 4 hours post-dose | 3.77 (NA) — N/A : not enough participants to calculate the standard deviation | 8.12 (2.36) |  |

27. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 1
Description: as for outcome 26
Time Frame: Week 1, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 1 | 5 | 1 | 2
ng/mL | 10.9 (NA) — N/A : not enough participants to calculate the standard deviation | 10.5 (6.57) | 21.3 (NA) — N/A : not enough participants to calculate the standard deviation | 22.3 (14.2)

28. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 2
Description: as for outcome 26
Time Frame: Week 2
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 2 | 2 | 2 | 2
ng/mL
  Week 2: 0.75 hour post-dose | 3.89 (2.76) | 3.69 (3.3) | 33.1 (19.2) | 34.9 (34.6)
  Week 2: 2 hours post-dose | 8.93 (2.36) | 14.3 (7.64) | 21.3 (4.53) | 33.6 (8.84)
  Week 2: 4 hours post-dose: number analyzed (Participants) | 2 | 1 | 2 | 2
  Week 2: 4 hours post-dose | 7.01 (2.69) | 11.1 (NA) — N/A : not enough participants to calculate the standard deviation | 13.6 (3.89) | 29.2 (0.354)

29. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 3
Description: as for outcome 26
Time Frame: Week 3, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 4 | 1 | 1 | 2
ng/mL | 7.09 (2.07) | 7.62 (NA) — N/A : not enough participants to calculate the standard deviation | 23.2 (NA) — N/A : not enough participants to calculate the standard deviation | 37.8 (0.849)

30. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 4
Description: as for outcome 26
Time Frame: Week 4, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 4 | 2 | 0 | 2
ng/mL | 4.08 (2.61) | 9.91 (3.53) |  | 24.0 (21.00)

31. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 6
Description: as for outcome 26
Time Frame: Week 6, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 4 | 2 | 0 | 1
ng/mL | 6.74 (2.42) | 12.7 (9.08) |  | 31.7 (NA) — N/A : not enough participants to calculate the standard deviation

32. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 8
Description: as for outcome 26
Time Frame: Week 8, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 5 | 1 | 0 | 0
ng/mL | 3.35 (2.75) | 13.9 (NA) — N/A : not enough participants to calculate the standard deviation |  |

33. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 10
Description: as for outcome 26
Time Frame: Week 10, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 4 | 2 | 0 | 0
ng/mL | 4.73 (1.26) | 11.3 (4.57) |  |

34. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 12
Description: as for outcome 26
Time Frame: Week 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 2 | 1 | 0 | 0
ng/mL
  Week 12: 0.75 hour post-dose | 0.382 (0.171) | 3.1 (NA) — N/A : not enough participants to calculate the standard deviation |  |
  Week 12: 2 hours post-dose | 4.62 (2.51) | 9.98 (NA) — N/A : not enough participants to calculate the standard deviation |  |
  Week 12: 4 hours post-dose | 3.58 (2.3) | 6.57 (NA) — N/A : not enough participants to calculate the standard deviation |  |

35. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 16
Description: as for outcome 26
Time Frame: Week 16, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 2 | 0 | 0 | 0
ng/mL | 5.71 (1.33) |  |  |

36. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 20
Description: as for outcome 26
Time Frame: Week 20, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 1 | 0 | 0 | 0
ng/mL | 0.794 (NA) — N/A : not enough participants to calculate the standard deviation |  |  |

37. Secondary Outcome: Plasma Concentrations of Osilodrostat (LCI699) at Week 24
Description: as for outcome 26
Time Frame: Week 24, 2 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Osilodrostat 1mg | Osilodrostat 2mg | Osilodrostat 3mg | Osilodrostat 5mg
Number analyzed (Participants) | 2 | 0 | 0 | 0
ng/mL | 6.51 (2.14) |  |  |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 68.0 weeks.
Description: AE description; Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Osilodrostat
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=9)
Myocardial infarction (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Pneumonia (Infections and infestations) | 1
Psychiatric symptom (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 5
Steroid withdrawal syndrome (Endocrine disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 3
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Reactive psychosis (Psychiatric disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Peripheral coldness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT02468193/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT02468193/SAP_001.pdf